CLINICAL TRIAL: NCT01786837
Title: A Prospective Trial to Study Whether Functional Magnetic Stimulation Enhances Gastrointestinal Motility in Patients With Chronic Constipation
Brief Title: Functional Magnetic Stimulation Enhances Gastrointestinal Motility in Patients With Chronic Constipation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-182; W81XWH-11-1-0707 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Constipation
Keywords: constipation; gastric emptying
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): FMS will be administered for 5 weeks
  Interventions: Device: Functional Magnetic Stimulation
- Sham (Sham Comparator): FMS at 5% intensity for 5 weeks
  Interventions: Device: Functional Magnetic Stimulation

INTERVENTIONS:
Device: Functional Magnetic Stimulation — 20 minute stimulation will be applied 5 days a week for 5 weeks
  Other Names: Commericially available magnetic stimulations with round magnetic coils.

SUMMARY:
The purpose of this study is to evaluate the effects of Functional Magnetic stimulation (FMS) on gastrointestinal motility in patients suffering from chronic constipation due to non-neurological issues.

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate the usefulness of FMS as a noninvasive method to stimulate the GI motility in individuals with non-neurological constipation by adopting a 5-week conditioning protocol performed in a hospital outpatient setting. FMS has demonstrated the ability to generate significant rectal pressure and enhance GI transit in normal and spinal cord injury subjects. With proper abdominal muscle conditioning, FMS may improve colonic motility partly due to improved abdominal muscle tone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* constipation defined by the Rome II criteria

Exclusion Criteria:

* Past history of abdominal surgery
* past history of diabetes mellitus
* past history of hypothyroidism
* past history of inflammatory bowel disease
* past history of significant psychiatric disturbances
* past history of drug abuse
* past history of cardiac pacemakers
* past history of metal implants
* patients who cannot travel to keep the follow up
* patients who are prisoners
* patients who are mentally handicapped
* patients who are pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of FMS in accelerating the gastric emptying in patients with non-neurological constipation after 5-week conditioning protocol | 5 weeks after conditioning

SECONDARY OUTCOMES:
Effectiveness of FMS in reducing the colonic transit time in patients with non-neurological constipation after a 5 week conditioning period | 5 weeks after conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Massarat Zutshi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Digestive Disease Institute, Cleveland, Ohio, United States